CLINICAL TRIAL: NCT03073694
Title: Phase II Single-Blind Randomized Trial Comparing Morbidity of Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy (CRS-HIPEC) Using Mitomycin-C Versus Melphalan for Colorectal Peritoneal Carcinomatosis
Brief Title: Comparing Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy (CRS-HIPEC) Using Mitomycin-C Versus Melphalan for Colorectal Peritoneal Carcinomatosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIT-2016-MAGIMelphVMitCHIPEC
Record Dates: First submitted 2017-02-09; First posted 2017-03-08 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Cancer, Appendiceal; ColoRectal Cancer
Keywords: Peritoneal Surface Disease; mitomycin-c; melphalan; Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy (CRS-HIPEC); Peritoneal Carcinomatosis
MeSH Terms: conditions — Appendiceal Neoplasms; Colorectal Neoplasms; Peritoneal Neoplasms | interventions — Mitomycin; Melphalan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mitomycin C Group (Active Comparator): Mitomycin-C initial dose of 15 mg/m2 (milligrams per meter squared) 45 minutes into the perfusion, a maintenance dose of 5 mg/m2 will be administered.
  Interventions: Drug: Mitomycin c
- Melphalan Group (Experimental): Melphalan 60 mg/m2 (milligrams per meter squared) 45 minutes into the perfusion.
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Mitomycin c — Mitomycin-c will be given to participants in Treatment Arm 1 as a one-time, intraoperative, intravenous administration for a duration of 90 minutes. 45 minutes into the perfusion, a maintenance dose will be administered.
  Other Names: Mutamycin; MTC
  Arms: Mitomycin C Group
Drug: Melphalan — Melphalan will be given to participants in Treatment Arm 2 as a one-time, intraoperative, intravenous administration for a duration of 90 minutes.
  Other Names: Alkeran
  Arms: Melphalan Group

SUMMARY:
The purpose of this trial is to compare the morbidity and mortality of CRS-HIPEC using mitomycin-C versus melphalan for colorectal peritoneal carcinomatosis. Morbidity and mortality will measured using the Comprehensive Complication Index (CCI) score, Common terminology criteria for adverse events (CTCAE version 4.03), and the Clavien-Dindo Classification.

DETAILED DESCRIPTION:
BACKGROUND: Peritoneal dissemination of cancer (peritoneal carcinomatosis) from gastrointestinal malignancies, meaning tumor deposits along the inside abdominal or pelvic wall and surfaces of the intestines and organs, has historically been considered a terminal disease. Although peritoneal surface tumors can respond to systemic therapy as a sole form of treatment, patient survival remains poor and cure is considered impossible.

A plasma-peritoneal barrier makes systemic therapy relatively ineffective against peritoneal surface disease. In the 1990's, cytoreductive surgery and hyperthermic intraperitoneal therapy (CRS-HIPEC) began to be popularized as a more effective treatment.

Hyperthermic intraperitoneal chemotherapy has several advantages. High-dose chemotherapy can be used due to the plasma-peritoneal barrier resulting in little absorption into the blood stream. Hyperthermia itself has cytotoxic effects and can increase the depth of tumor penetration by the chemotherapeutic agent up to 3 mm and moreover can potentiate its antineoplastic effects. Although CRS-HIPEC has been considered standard treatment for ruptured appendiceal neoplasms and primary peritoneal mesothelioma, in the past decade its indications have broadened to other peritoneal surface malignant processes.

Historically, morbidity and mortality associated with CRS-HIPEC was considerably higher than other complex operations, and thus its use was often discouraged. However, in recent times, especially in high-volume centers, morbidity and mortality has drastically improved. Due to recent improvements in mortality after major surgical interventions, including HIPEC, the focus has shifted toward other endpoints besides efficacy, such as morbidity, quality of life and cost.

While HIPEC is universally felt to be a vital component after cytoreductive surgery, there is a lack of consensus on the optimal regimen, especially the chemotherapeutic agent that should be used. In the United States, the most commonly used agent during HIPEC is mitomycin-C, however, it remains unknown if mitomycin-C is the optimal drug to use with regards to toxicity and survival.

Randomized prospective studies are needed comparing the toxicity and effectiveness of HIPEC with mitomycin-C to other agents.

OBJECTIVE: To compare morbidity and mortality after CRS-HIPEC utilizing mitomycin-C versus melphalan.

METHODS: In this study, patients will be randomized to one of two treatment arms: Arm 1.) Mitomycin-C initial dose of 15 mg/m2, 45 minutes into the perfusion a maintenance dose of 5 mg/m2 will be administered; or Arm 2): Melphalan 60 mg/m2 45 minutes into the perfusion. Morbidity will be measured during immediate and short-term surgical recovery (up to 90 days post-hospital discharge). Mortality will be measured beginning with the date of surgery and ending with the date of participant death.

ELIGIBILITY:
Inclusion Criteria

* Ability to understand and the willingness to sign a written informed consent.
* Peritoneal Surface Disease (PSD) due to Colorectal Cancer or High-Grade Appendiceal Cancer
* No clear evidence of systemic metastases
* No prior CRS-HIPEC treatment
* Patient has a planned CC0 (Complete Macroscopic Cytoreduction (visual)) cytoreduction - NOTE: randomization occurs during surgery and not before; if, during surgery, the PI/SubI discerns that all disease cannot be removed surgically, the participant will be considered a "screen failure", HIPEC will not be performed, and the participant will be removed from the study. If participant is removed from the study, PI / surgeon will decide if standard of care surgery will proceed.
* Age 18 - 75
* ECOG (Eastern Cooperative Oncology Group) Score 0 - 2
* Recorded ASA (American Society of Anesthesiologist Classification) classification - as determined by the anesthesiologist (particular value not required - only recording of the classification is required).
* Medically fit to undergo complex major abdominal surgery, as determined by examination by PI / Sub-Is.
* Medically fit to receive systemic chemotherapy, as determined by examination by PI / Sub-Is.
* Adequate organ and marrow function as defined below:

  * leukocytes ≥ 3,000/mcL (microliter)
  * absolute neutrophil count ≥ 1,500/mcL
  * platelets ≥ 100,000/mcL
  * total bilirubin within normal institutional limits
  * AST (Aspartate aminotransferase) (SGOT [Serum Glutamic Oxaloacetic Transaminase]) ≤ 2.5 X institutional upper limit of normal
  * ALT (Alanine Aminotransferase) (SPGT [Serum Glutamic Pyruvic Transaminase]) ≤ 2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

  * A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
  * Men of child-bearing potential must not donate sperm while on this study and for 90 days after the study treatment (surgery with HIPEC).

Exclusion Criteria Participants meeting any of the exclusion criteria at baseline will be excluded from study participation.

* Current or anticipated use of other investigational agents while participating in this study.
* Patient has received systemic chemotherapy or radiotherapy within 4 weeks prior to study enrollment.
* Patient has not recovered sufficiently (PI will judge patient recovery status) from adverse events due to agents administered more than 4 weeks prior to enrollment on this study.
* Patient has history of or currently has non-peritoneal surface metastatic disease in addition to peritoneal surface malignancy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to mitomycin-C or melphalan.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, life-threatening cardiac arrhythmia, severe pulmonary disease, uncontrolled diabetes, severe kidney disease or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing. There is a potential for congenital abnormalities and for this regimen to harm nursing infants.
* Patient actively being treated for other malignancy (current active treatment of early stage squamous or basal cell carcinomas of the skin is allowed, excluding treatment with other investigational agents and systemic chemotherapy or radiotherapy).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07-14 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Complication Index (CCI) score. | Every 3 months until Year 2
  CCI will be evaluated using the following data: morbidity, mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Mazin Al-kasspooles, MD, Principal Investigator — The University of Kansas - Cancer Center
Locations (1):
- The University of Kansas Medical Center, Westwood, Kansas, United States

IPD SHARING:
Plan to Share IPD: No